CLINICAL TRIAL: NCT06833190
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of a Multiple Dose Regimen of REGN5381, an NPR1 Monoclonal Antibody Agonist, in Participants With Uncontrolled Hypertension
Brief Title: REGN5381 in Adult Participants With Uncontrolled Hypertension
Acronym: NATRIX-SBP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R5381-UHTN-2410
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Uncontrolled Hypertension
Keywords: High blood pressure; Systolic Blood Pressure (SBP)
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- REGN5381 Low Dose (Experimental): Randomized as described in the protocol
  Interventions: Drug: REGN5381
- REGN5381 High Dose (Experimental): Randomized as described in the protocol
  Interventions: Drug: REGN5381
- Placebo (Placebo Comparator): Randomized as described in the protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN5381 — Administered per the protocol
  Arms: REGN5381 High Dose; REGN5381 Low Dose
Drug: Placebo — Administered per the protocol
  Arms: Placebo

SUMMARY:
This study is researching an experimental drug called REGN5381 (called "study drug"). The study is focused on uncontrolled hypertension (high blood pressure despite being on one or more antihypertensive drugs).

The aim of the study is to see how effective the study drug is in reducing blood pressure. The study is designed as a 2-part study with participants initially enrolling in Part A. Part B of the study will commence and enroll the remaining study participants.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

DETAILED DESCRIPTION:
As of October 15, 2025, this study has been terminated, and all future onsite visits have been canceled. However, participants have been asked to report safety information to the trial helpline until January 15, 2026.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adults with SBP ≥130 mm Hg and SBP ≤180 mm Hg at both screening and randomization visit, as described in the protocol
2. ≥ 40 and ≤85 years on a stable regimen of ≥1 anti-hypertensive therapy for at least 1 month at the time of screening or ≥30 and <40 years on a stable regimen of ≥3 anti-hypertensive therapies for at least 1 month at the time of screening

Key Exclusion Criteria

1. Heart rate >100 bpm as described in the protocol
2. Body mass index >45 kg/m2 as described in the protocol
3. Glomerular filtration rate (GFR) <30 mL/min/1.73m2 at screening as described in the protocol
4. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≥3x upper limit of normal (ULN) as described in the protocol

NOTE: Other protocol-defined Inclusion/Exclusion Criteria apply

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Unattended Automated Office-Based Blood Pressure (AOBP) Systolic Blood Pressure (SBP) | At week 12

SECONDARY OUTCOMES:
Unattended AOBP SBP in stage 3 Chronic Kidney Disease (CKD) participants | At week 12
Unattended AOBP SBP in participants on ≥3 anti-hypertensive therapies | At week 12
Time-weighted average AOBP SBP | Through week 12
Time-weighted average AOBP Diastolic Blood Pressure (DBP) | Through week 12
AOBP SBP | From baseline to weeks 2, 4 and 8
AOBP DBP | From baseline to weeks 2, 4, 8 and 12
Mean SBP by 24-hour Ambulatory Blood Pressure Monitoring (ABPM) | At week 12
Concentrations of REGN5381 in serum | Through week 20
Occurrence of Treatment Emergent Adverse Events (TEAEs) | Up to week 23
Severity of TEAEs | Up to week 23
Occurrence of TEAEs leading to discontinuation of study drug | Up to week 23
Occurrence of Anti-Drug Antibodies (ADAs) to REGN5381 | Through week 20
Titer of ADAs to REGN5381 | Through week 20

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- United Kingdom (3):
  - Protas, Car Park of Asda Huyton Supercentre, Huyton, Liverpool
  - Protas, Two New Bailey Square, Salford, Manchester
  - Protas, Car Park of Asda Pilsworth Road, Bury

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/